CLINICAL TRIAL: NCT00517387
Title: The Effects of Quetiapine XR on Cognition, Mood and Anxiety Symptoms in SSRI-Resistant Unipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Dr. Allan Young, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H07-00629
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Unipolar Depression
Keywords: Depression; SSRI; Atypical Antipsychotic; Cognition; Mood; Quality of Life
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): All patients will receive Quetiapine XR at an initial dose of 50mg/day to be increased incrementally (dose of 50mg/day 2 and 150mg/day 3) to achieve a target dose of 300 mg/day by day 4. Tablets will be self-administered early each night.
  Interventions: Drug: Quetiapine XR

INTERVENTIONS:
Drug: Quetiapine XR — All patients will receive Quetiapine XR at an initial dose of 50mg/day to be increased incrementally (dose of 50mg/day 2 and 150mg/day 3) to achieve a target dose of 300 mg/day by day 4. Tablets will be self-administered early each night.

SUMMARY:
Recently published work has examined the effects of "atypical antipsychotics" in SSRI-treatment resistant patients. In these studies, patients with unipolar depression who were treated with SSRI's, but not responsive to treatment after 4 or more weeks, were supplemented with an atypical. The atypical antipsychotics were found to diminish depression symptoms, as well as benefit sleep quality.

We propose a similar study with Quetiapine XR, focusing on thinking processes, mood and anxiety. Patients with depression who are SSRI treatment resistant will be treated with Quetiapine. Cognition will be evaluated in the UBC Mood Disorders Clinic two times: first before Quetiapine addition, then after 8 weeks. Depression symptoms and other measurements will be done at the 9 time points: before Quetiapine, and each week after treatment has begun.

The primary purpose of this study is to evaluate the superiority of Quetiapine XR compared to placebo as augmentation therapy in treatment of anxiety and depressive symptoms in SSRI-nonresponsive unipolar patients. Secondarily, we would like to evaluate the safety and tolerability of quetiapine as augmentation therapy in SSRI-nonresponsive unipolar patients.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled study, in which patients will receive treatment of Quetiapine XR for 8 weeks. All patients will receive Quetiapine XR at an initial dose of 50mg/day to be increased incrementally (dose of 50mg/day 2 and 150mg/day 3) to achieve a target dose of 300 mg/day by day 4. Tablets will be self-administered early each night. Patient's results will be compared to their own baseline measurements, in a double-blind fashion.

Recruited patients will be evaluated at nine time points: a baseline prior to treatment (t = -7 days), an assessment one week after treatment has begun (t = 7 days), two weeks after (t = 14 days), three weeks after (t = 21 days), four weeks after (t = 28 days), five weeks after (t = 35 days), six weeks after (t = 42 days), seven weeks after (t = 49 days) and after 8 weeks of treatment (t = 56 days). Evaluation of cognition, mood and anxiety, will be done blind to which time point is being measured.

Basic blood work (fasting blood glucose, lipid screen including triglycerides, urea and electrolytes, cytokines and neuroimmune markers) will performed on each patient both at baseline (t = -7 days) and at t = 56 days. At 4 weeks, blood sample will be taken for fasting plasma glucose, HbA1c and transaminases. At baseline (-7 days) and completion (56 days) a battery of neurocognitive-impairment tests (see Appendix A) will be administered. In addition, the Hamilton Rating Scale for Depression (21-ITEM HAM-D GRID), Montgomery -Asberg Depression Rating Scale (MADRS), Hamilton Ratings Scale for Anxiety (HAM-A), the UKU Side Effect Rating Scale, and the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) will also be assessed by the research team.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. A diagnosis of Unipolar Depression by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV-TR)
3. Females and males aged 19-65 years
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment
5. Able to understand and comply with the requirements of the study
6. Minimum 21-item HAM-D GRID score of 15
7. Prior treatment with therapeutic doses of an SSRI-type antidepressant for at least 6 weeks
8. Unsatisfactory response to treatment, as determined by clinician, for at least 6 weeks.

Exclusion Criteria:

1. Pregnancy or lactation
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria
3. English as a second language
4. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
5. Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
6. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
7. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
8. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
9. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
10. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
11. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
12. Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
13. Involvement in the planning and conduct of the study
14. Previous enrolment or randomisation of treatment in the present study.
15. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
16. Previous head injury, associated with loss of consciousness.
17. Neurological disorder.
18. Significant physical health problem
19. An absolute neutrophil count (ANC) of 1.5 x 109 per liter;
20. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM defined as enrollment glycosylated hemoglobin (HbA1c) >8.5%.
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
    * Not under physician care for DM
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
    * Physician responsible for patient's DM care has not approved patient's participation in the study. Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomization. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks.
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome will be measurements of cognitive function, determined both prior to treatment and after 8 weeks of treatment. | 8 weeks

SECONDARY OUTCOMES:
To evaluate Quetiapine XR compared to placebo, in SSRI-nonresponsive unipolar patients, in treatment of anxiety and depressive symptoms and biomarkers, improving patient's overall quality of life, and to evaluate its safety and tolerability. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allan Young, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Hospital, Vancouver, British Columbia, Canada